CLINICAL TRIAL: NCT06230601
Title: Effect of Cough Trick Method and Pinwheel Blowing in Blood Collection in School-Age Children on the Level of Pain: Randomized Controlled Study
Brief Title: Effect of Cough Trick Method and Pinwheel Blowing in Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Özlem Selime MERTER, ASSISTANT PROFESSOR, Firat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/ 01-50
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Child Development; Nursing Care; Pain
Keywords: children; nurse; blood collection; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group (Experimental): cough trick method will be used in the blood collection process from the children in the experimental group.
  Interventions: Other: Cough Trick Method
- Active comprator (Active Comparator): Pinwheel Blowing method will be used in the blood collection process from the children in the experimental group.
  Interventions: Other: Pinwheel Blowing method
- control group (No Intervention): Routine application of the unit will be made

INTERVENTIONS:
Other: Cough Trick Method — During the Blood Collection Procedure in School-Age Children, one group will use the Cough Trick Method
  Other Names: Pinwheel Blowing Method
  Arms: experimental group
Other: Pinwheel Blowing method — Pinwheel Blowing method
  Arms: Active comprator

SUMMARY:
This study aimed to examine the effect of the cough trick method and pinwheel blowing on the severity of pain during blood collection in school-age children.The study will be conducted with children aged 6-12 years who are subjected to blood tests by a pediatrician."Descriptive Questionnaire", "Visual Analogue Scale (VAS)", "FLACC Pain Rating Scale" and "Wong-Baker Faces Pain Rating Scale (WBFPRS)" will be used to collect data.The data will be uploaded to the computer and coded by the researchers, and the data will be evaluated in the SPSS package program.The sociodemographic data of the children participating in the study will be given as numbers and percentage distributions. Appropriate tests will be used by analyzing the data for normal distribution. The statistical significance level of the study was determined as p< 0.05. In addition, at the end of the research, the status of working with sufficient sample size will be tested with post-hoc power analysis.

DETAILED DESCRIPTION:
Purpose of the study: This study aimed to examine the effect of the cough trick method and pinwheel blowing on the severity of pain during blood collection in school-age children.

Type of Study: It is a randomized controlled study.

Location and Characteristics of the Study: It will be conducted in the pediatric blood collection unit of Fırat University Hospital, with children aged 6-12 who are subjected to blood tests by a pediatrician.

Population-Sample: The population of the study will consist of children who applied for blood collection in the pediatric blood collection unit of Fırat University Hospital. A pilot study will be conducted to determine the number of samples. For the pilot study, 20 participants will be taken from each group and a total of 60 samples will be taken. As a result of the pilot study, power analysis will be performed and the number of samples will be determined. Randomization will be done to assign the participants to the groups. Grouping will be done using simple random sampling. Randomization will be provided using the Random Sequence Generator on the www.random.org website. Each participant who volunteers to participate in the study and meets the criteria will be given a number. Accordingly, which number will take place in which group will be determined in advance.

Data collection tools: Questionnaire", "Visual Analogue Scale (VAS)", "FLACC Pain Rating Scale" and "Wong-Baker Faces Pain Rating Scale (WBFPRS)" will be used to collect data.

Data Collection: The research will be carried out in three stages. Stage 1: Groups of parent-child pairs who come to the blood collection unit, voluntarily participate in the research, and meet the inclusion criteria will be determined in line with the randomization method within the scope of the research. Study data will be collected in 3 groups. Two groups will be the intervention group and the third group will be the control group.

Group 1: cough trick group 2nd group is the pinwheel blower group. Group 3 will constitute the control group. Stage 2: Information about the children assigned to the groups will be obtained using the "Introductory Question Form".

Stage 3: Blood collection will be performed by the same nurse (a volunteer nurse with 5 years of experience in pediatric blood collection) to eliminate differences that may occur due to nurse differences. Blood samples from children will be taken with a 21 gauge x 1.5 inch vacuum blood collection needle. It will be ensured that the parent accompanies the child throughout all procedures.

Pain intensity will be measured through observation and physiological responses of the child, parent, and nurse. The child's pain intensity will be rated by the parent, the nurse (a pediatric nurse with 5 years of experience, independent of the blood draw) and the child himself before and after the blood draw. To determine pain severity, parents will use VAS, the nurse will use FLACC, and the child will use FACES scale.

Heart rate is the physiological measure used to report pain intensity, and the heart rate of the children in the study will be recorded before and after the procedure using a pulse oximeter device at 2-minute intervals. The demographic questionnaire will be filled out by the children's parents 10 minutes before the procedure.

The statistical significance level of the study was determined as p< 0.05. In addition, at the end of the research, the status of working with sufficient sample size will be tested with post-hoc power analysis.

ELIGIBILITY:
Inclusion Criteria:

* School age children ages 6-12.
* Peripheral intravenous catheter (PIC) application was performed by the same nurse (with at least 5 years of experience).
* Able to express himself/herself verbally
* No visual or auditory problems

Exclusion Criteria:

* Children who received tropical anesthetic before the procedure
* Children whose first attempt to draw blood was unsuccessful
* Children who have taken analgesic medication within 24 hours before blood sampling
* Children with a body temperature of 37.5 ºC and above, mental or neurological disorders, a medical history of fainting or chronic diseases requiring frequent blood sampling, and those who have previously undergone surgery will be excluded from the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Scale | 1 day
  This method, which is aimed at determining the severity of pain, aims to explain the patient's pain in numbers. Absence of pain (0) is evaluated as unbearable pain (10) on numerical scales.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep KİSECİK ŞENGÜL, Study Chair — Kirikkale Universty; Rüveyda OĞUZ, Study Chair — Firat University
Locations (1):
- Fırat Univesity, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merter OS, Sengul ZK, Oguz R. Effects of blowing pinwheel and cough trick on pain in 6- to 12-year-old children during venipuncture: A randomized controlled trial. J Pediatr Nurs. 2025 Jul-Aug;83:30-37. doi: 10.1016/j.pedn.2025.04.023. Epub 2025 Apr 24. PMID 40279824